CLINICAL TRIAL: NCT06389643
Title: Comparison of Safety and Efficacy of Four-Point Scleral Intraocular Lens Fixation and Yamane Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Military Institute od Medicine National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/WIM/2021
Record Dates: First submitted 2024-04-17; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Aphakia
Keywords: scleral fixation IOL; sutureless fixation IOL; four-point scleral fixation; Yamane technique; aphakia
MeSH Terms: conditions — Aphakia

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Four-point scleral fixation group (Active Comparator): Four-point scleral fixation group
  Interventions: Procedure: Four-point scleral fixation of Akreos AO60 IOL
- Yamane technique group (Active Comparator): Yamane technique group
  Interventions: Procedure: Sutureless scleral fixation of AcrySof MA60AC IOL with Yamane technique

INTERVENTIONS:
Procedure: Four-point scleral fixation of Akreos AO60 IOL — Intrascleral tunnels were marked at a distance of 2 mm from the corneal limbus, 6 mm apart (4 in number) after retrobulbar anesthesia. Next corneal incisions were performed. An artificial lens was then implanted into the anterior chamber. The 6-0 polypropylene suture was introduced into the anterior chamber through openings in the cornea. The next stage was to perform a sclerotomy using a 30G needle. Then the needle was passed through the hole in the haptic and 6-0 polypropylene suture was inserted into the needle hole and guided outside. The other end of the suture, passed through the opening in the haptic, was placed in the lumen of the needle and carried out through another sclerotomy and then externalised. This maneuver was repeated with another haptics as well. Correct position of the IOL in the eye was achieved by pulling on the ends of the monofilament. The ends of sutures were trimmed and cauterized. The melted tips of the sutures were then fixed subconjunctivally.
  Arms: Four-point scleral fixation group
Procedure: Sutureless scleral fixation of AcrySof MA60AC IOL with Yamane technique — The surgery was performed under retrobulbar anesthesia. The first step of the procedure was to mark the locations of the intrascleral tunnels (2 mm from the corneal limbus) and locate them at a distance of 180° from each other to prevent the lens from tilting in the eyeball. Openings in the cornea were done. Three-piece IOL was implanted into the anterior chamber. The first sclerotomy was performed through the conjunctiva using a 30G needle 2 mm from the limbus. One of the haptics was inserted into the needle lumen and then brought out. Same procedure was performed with another haptic at a distance of 180°. The next step was to perform cautery of the tips of the haptics, obtaining a 0.3 mm collar that prevents the risk of the haptic coming out of the tunnel and displacing the lens inside the eyeball. The tips of the haptics were finally gently inserted into the scleral canals and covered with conjunctiva.
  Arms: Yamane technique group

SUMMARY:
Comparison of safety and efficacy of two scleral fixation intraocular lens (IOL) methods of four-point scleral fixation ( Akreos AO60) and the Yamane technique (AcrySof MA60AC)

DETAILED DESCRIPTION:
Purpose of the study is to compare two methods of scleral fixation of IOL: two-point fixation of AcrySof MA60AC IOL (Alcon) using Yamane technique and four-point fixation of the Akreos AO60 IOL (Bausch & Lomb) using polypropylene suture. The investigators rated the BCVA, refractive outcomes, intraocular pressure, and also determined intra- and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* only adult men and women with aphakia without capsular support

Exclusion Criteria:

* Fuchs' dystrophy
* corneal haze or scarring
* history of corneal transplantation
* astigmatism of more than 2,0D
* clinically active uveitis
* advanced glaucoma
* macular diseases that affect visual acuity (age-related macular degeneration, diabetic maculopathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
BCVA | before and 12 months after surgery
  The change of best- corrected visual acuity
RE | 12 months after surgery
  Postoperative total refractive error
ECC | before and 12 months after surgery
  corneal endothelial cell density

SECONDARY OUTCOMES:
Number of complications | from day 1 until 12 months after surgery
  Rate of complications

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Blagun, MD, Principal Investigator — Military Institute of Medicine National Research Institute
Locations (1):
- Military Institute of Medicine - National Research Institute, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blagun N, Krix-Jachym K, Rekas M. Comparison of Safety and Efficacy of Four-Point Scleral Intraocular Lens Fixation and the Yamane Technique. Ophthalmol Ther. 2024 Jul;13(7):1955-1966. doi: 10.1007/s40123-024-00962-7. Epub 2024 May 21. PMID 38771460